CLINICAL TRIAL: NCT05013684
Title: Benign Paroxysmal Positional Vertigo in Older Adults: Treatment Efficacy and the Impact on Balance, Inactivity and Frailty
Brief Title: Benign Paroxysmal Positional Vertigo in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, JSpildooren, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPPVOA-001
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older adults with BPPV (Active Comparator)
  Interventions: Other: Particle Repositioning Maneuver
- Older adults without BPPV (No Intervention)

INTERVENTIONS:
Other: Particle Repositioning Maneuver — treatment with Particle Repositioning Maneuver
  Arms: Older adults with BPPV

SUMMARY:
Despite the growing research on Benign Paroxysmal Positioning Vertigo (BPPV), the impact and treatment efficacy on balance, physical activity (and consequently) frailty in elderly is lacking. Also, the added value of the video Head Impulse Test (vHIT) in this population has never been studied before. With insights gained from this research, we hope to contribute to an efficient treatment of BPPV in this growing population and to minimize its impact and healthcare burden.

ELIGIBILITY:
Inclusion Criteria:

* Persons ≥ 65 years old
* Able to stand independent for at least 30 seconds
* Able to walk (with or without) walking aid for at least 10 meters
* Patients diagnosed with posterior semicircular canal BPPV
* Patients diagnosed with lateral-semicircular canal BPPV

Exclusion Criteria:

* Unable to understand and follow simple instructions (e.g. due to severe dementia, hearing loss or visual impairment)
* Persons temporarily or permanently living in a residential or psychiatric care centre, a home for the disabled or rehabilitation centre
* Persons with contra-indications for the diagnostic maneuver, vHIT or caloric irrigation test (e.g. severe limitation in mobility of the cervical spine of perforation of the tympanic membrane)
* Persons with other (acute) vestibular disorders and who as a result no longer meet the above mentioned diagnostic criteria for BPPV
* Persons with evolutionary disorders of the central nervous system (e.g. multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis).
* Persons who are already taking antivertigo drugs.
* Persons still in the rehabilitation phase after an orthopedic or cardiovascular incident.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The mini Balance Evalutation System test (miniBEStest) | baseline
  The MiniBEStest is a 14-item test that measures 4 different balance control systems: anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. Items are scored on a 3-level ordinal scale.
  The CTSIB is used to assess sensory contributions to postural control during 6 sensory conditions: stand on firm surface with eyes open, stand on foam surface with eyes open, stand on firm surface with visual conflict dome, stand on foam surface with visual conflict dome, stand on firm surface with eyes closed and stand on foam surface with eyes closed.
The mini Balance Evalutation System test (miniBEStest) | month 1
  The MiniBEStest is a 14-item test that measures 4 different balance control systems: anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. Items are scored on a 3-level ordinal scale.
  The CTSIB is used to assess sensory contributions to postural control during 6 sensory conditions: stand on firm surface with eyes open, stand on foam surface with eyes open, stand on firm surface with visual conflict dome, stand on foam surface with visual conflict dome, stand on firm surface with eyes closed and stand on foam surface with eyes closed.
The mini Balance Evalutation System test (miniBEStest) | month 3
  The MiniBEStest is a 14-item test that measures 4 different balance control systems: anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. Items are scored on a 3-level ordinal scale.
  The CTSIB is used to assess sensory contributions to postural control during 6 sensory conditions: stand on firm surface with eyes open, stand on foam surface with eyes open, stand on firm surface with visual conflict dome, stand on foam surface with visual conflict dome, stand on firm surface with eyes closed and stand on foam surface with eyes closed.
The mini Balance Evalutation System test (miniBEStest) | month 6
  The MiniBEStest is a 14-item test that measures 4 different balance control systems: anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. Items are scored on a 3-level ordinal scale.
  The CTSIB is used to assess sensory contributions to postural control during 6 sensory conditions: stand on firm surface with eyes open, stand on foam surface with eyes open, stand on firm surface with visual conflict dome, stand on foam surface with visual conflict dome, stand on firm surface with eyes closed and stand on foam surface with eyes closed.
10 meter walk test | Baseline
  During the 10 meter walk test the participant is instructed to walk 10 meter at his/her preferred walking speed. Gait parameters will be assessed.
10 meter walk test | month 1
  During the 10 meter walk test the participant is instructed to walk 10 meter at his/her preferred walking speed. Gait parameters will be assessed.
10 meter walk test | month 3
  During the 10 meter walk test the participant is instructed to walk 10 meter at his/her preferred walking speed. Gait parameters will be assessed.
10 meter walk test | month 6
  During the 10 meter walk test the participant is instructed to walk 10 meter at his/her preferred walking speed. Gait parameters will be assessed.
physical activity level measurde by an accelerometer (MOX) | baseline
  Objective measurement of physical activity level of four days will be done by an accelerometer (MOX), that measures time spent in certain positions. The accelerometer is attached to the upper leg of the participant.
physical activity level measurde by an accelerometer (MOX) | month 1
  Objective measurement of physical activity level of four days will be done by an accelerometer (MOX), that measures time spent in certain positions. The accelerometer is attached to the upper leg of the participant.
physical activity level measurde by an accelerometer (MOX) | month 3
  Objective measurement of physical activity level of four days will be done by an accelerometer (MOX), that measures time spent in certain positions. The accelerometer is attached to the upper leg of the participant.
physical activity level measurde by an accelerometer (MOX) | month 6
  Objective measurement of physical activity level of four days will be done by an accelerometer (MOX), that measures time spent in certain positions. The accelerometer is attached to the upper leg of the participant.
The International Physical Activity Questionnaire | Baseline
  used to measure the level of physical activity by questionnaire. This questionnaire consists of 31 questions divided over 5 subcategories. A higher score means a higher level of physical activity.
The International Physical Activity Questionnaire | Month 1
  used to measure the level of physical activity by questionnaire. This questionnaire consists of 31 questions divided over 5 subcategories. A higher score means a higher level of physical activity.
The International Physical Activity Questionnaire | Month 3
  used to measure the level of physical activity by questionnaire. This questionnaire consists of 31 questions divided over 5 subcategories. A higher score means a higher level of physical activity.
The International Physical Activity Questionnaire | Month 6
  used to measure the level of physical activity by questionnaire. This questionnaire consists of 31 questions divided over 5 subcategories. A higher score means a higher level of physical activity.
Frailty | baseline
  Frailty is defined as a clinical syndrome in which three or more of the following criteria are present: unintentional weight loss (more than 3 kg during last year and/or BMI ≤ 21 kg/m2), weakness (unable to rise from a chair), self-reported exhaustion, slow walking speed (velocity on 10 meter walk test) and low physical activity (answering 'no' to the question 'do you perform regular physical activity as walking, gardening or sport).
Frailty | month 1
  Frailty is defined as a clinical syndrome in which three or more of the following criteria are present: unintentional weight loss (more than 3 kg during last year and/or BMI ≤ 21 kg/m2), weakness (unable to rise from a chair), self-reported exhaustion, slow walking speed (velocity on 10 meter walk test) and low physical activity (answering 'no' to the question 'do you perform regular physical activity as walking, gardening or sport).
Frailty | month 3
  Frailty is defined as a clinical syndrome in which three or more of the following criteria are present: unintentional weight loss (more than 3 kg during last year and/or BMI ≤ 21 kg/m2), weakness (unable to rise from a chair), self-reported exhaustion, slow walking speed (velocity on 10 meter walk test) and low physical activity (answering 'no' to the question 'do you perform regular physical activity as walking, gardening or sport).
Frailty | month 6
  Frailty is defined as a clinical syndrome in which three or more of the following criteria are present: unintentional weight loss (more than 3 kg during last year and/or BMI ≤ 21 kg/m2), weakness (unable to rise from a chair), self-reported exhaustion, slow walking speed (velocity on 10 meter walk test) and low physical activity (answering 'no' to the question 'do you perform regular physical activity as walking, gardening or sport).

SECONDARY OUTCOMES:
the Montreal Cognitive Assessment (MOCA) | Baseline
  Cognitive function of older adults with BPPV will be compared to cognitive function of older adults without BPPV. Cognitive function will be assessed with the Montreal Cognitive Assessment (MOCA). MOCA assesses short term memory, visuospatial abilities, executive functions, attention and working memory, language and orientation to time and place.
the 15-item Geriatric Depression Scale | baseline
  Depressive feeling will be measured with the 15-item Geriatric Depression Scale
the 15-item Geriatric Depression Scale | Month 1
  Depressive feeling will be measured with the 15-item Geriatric Depression Scale
the 15-item Geriatric Depression Scale | Month 3
  Depressive feeling will be measured with the 15-item Geriatric Depression Scale
the 15-item Geriatric Depression Scale | Month 6
  Depressive feeling will be measured with the 15-item Geriatric Depression Scale
Age | Throug study completion, an average of 6 months
  Years
Height | Throug study completion, an average of 6 months
  meters
BPPV-symptomatology | Throug study completion, an average of 6 months
medication use | Throug study completion, an average of 6 months
  medication use will be questioned
Living situation | Throug study completion, an average of 6 months
  Living situation wil be questioned
Walking aid | Throug study completion, an average of 6 months
  Walking aid wil be questioned
Fall history | Up to the end of the study
  Fall History will be measured during the follow-up period by a 2-weekly telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Joke Spildooren, prof. dr., Principal Investigator — Hasselt University; Sara Pauwels, drs., Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium